CLINICAL TRIAL: NCT02120820
Title: An Evaluation of the Clinical Efficacy of Massage Therapy in a Multisensory Environment for Residents With Severe and Profound Intellectual Disabilities
Brief Title: Effect of Massage Therapy in a Multisensory Environment for Intellectual Disabilities
Acronym: MT-MSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Wai-Tong Chien, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HongKongPU
Record Dates: First submitted 2014-04-16; First posted 2014-04-23 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Behavior Disturbance; Muscle Hypotonia
Keywords: massage; multisensory environment; challenging behaviours; relaxation
MeSH Terms: conditions — Muscle Hypotonia | interventions — Massage; Manual Lymphatic Drainage; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Multisensory environment (Active Comparator): Multisensory environment (MSE): 30 minutes/session, twice a week for 10 weeks
  Interventions: Behavioral: Multisensory environment (MSE)
- Massage therapy (Active Comparator): Massage therapy (MT): 15 minutes/session, twice a week for 10 weeks
  Interventions: Behavioral: Massage therapy (MT)
- Control group (Other): Control group: usual care for 10 weeks, with attention and interactions with the caregivers only.
  Interventions: Other: Control group
- Massage in multisensory environment (Active Comparator): Participants receive 15 minutes massage therapy in multisensory environment (MT-MSE), twice a week for 10 weeks.
  Interventions: Behavioral: Multisensory environment (MSE); Behavioral: Massage therapy (MT); Behavioral: Massage therapy in multisensory environment (MT-MSE)

INTERVENTIONS:
Behavioral: Multisensory environment (MSE) — Participants are staying in multisensory environment (MSE only) for 30 minutes in each session, and twice per week for 10 weeks. An enabler stays with the participant throughout the session.
  Other Names: Sensory stimulation; Snoezelen
  Arms: Massage in multisensory environment; Multisensory environment
Behavioral: Massage therapy (MT) — A trained massage therapist provides 15 minutes massage therapy (MT) to the participants, twice a week for 10 weeks. The massage therapist acts as an enabler.
  Other Names: Massage; Manual massage
  Arms: Massage in multisensory environment; Massage therapy
Other: Control group — Usual residential care will be given to these participants. Only attention and social interactions from the enabler will be provided.
  Other Names: Placebo; no intervention
  Arms: Control group
Behavioral: Massage therapy in multisensory environment (MT-MSE) — Participants receive 15 minutes massage therapy while staying in multisensory environment for 30 minutes, twice a week for 10 weeks.
  Other Names: Massage; Sensory environment
  Arms: Massage in multisensory environment

SUMMARY:
The aim of this study is to evaluate the effectiveness of multisensory environment (MSE) and/or massage therapy (MT) in residents with severe and profound intellectual disabilities (ID) who received massage therapy in MSE, activities in MSE alone, massage therapy in usual care environment, or usual care with attention.

Since there has not yet been any conclusive evidence to show the clinical efficacy of MT and MSE on relaxation and reducing challenging behaviours, the following null hypotheses are suggested:

1. There will not be any differences on reducing heart and respiration rates between MT-MSE, MT, MSE, and usual care only over the 10-week intervention period and a 2-week follow-up.
2. There will not be any differences on adaptive behaviours and levels of alertness between MT-MSE, MT, MSE, and control group over the 10-week intervention period and a 2-week follow-up.
3. There will not be any differences on frequency and severity of challenging behaviours between MT-MSE, MT, MSE, and control group over the 10-week intervention period and a 2-week follow-up.

DETAILED DESCRIPTION:
Design:

This study adopts a mixed methods research design, in which both quantitative (i.e., randomized controlled trial design) and qualitative (exploratory) approaches will be used.

Methods:

After the study criteria are checked and met and proxy consent has been obtained, the participants will undergo a period of washout (4 weeks) from the current multisensory environment (MSE) and/or massage therapy (MT) sessions. After that, the baseline measurement of all outcome measures will be taken. All of them will then be randomly assigned to one of the four study groups, including three treatment groups, namely massage therapy in MSE (MT-MSE), MSE only and massage therapy in usual care environment (MT), and one control (routine care) group.

The effects of the three proposed interventions and routine care only groups on the study outcomes, including frequency and severity of challenging behaviour, adaptive behaviour, alertness level, and heart and respiration rate, will be compared between groups at baseline, interim (i.e., 5 weeks after the interventions started), immediately after completion of the interventions (i.e. 10 weeks after the interventions started), and 2 weeks follow up (i.e. at 12 weeks from the start of intervention, but no intervention at week 11 and 12). A pilot study will be conducted to review the feasibility and clarity of the study procedure, intervention protocols, and outcome measurements in around 30 patients with similar clinical characteristics (i.e., 8 subjects per groups) before starting the main study.

Primary outcomes of the study are frequency and severity of challenging behaviours, and the physiological signs (i.e., respiration and pulse rate). The secondary outcomes are the levels of alertness and adaptive behaviours.

Primary nurses who are responsible to formulate the individualized MSE and/or MT programs of the participants in the three treatment groups will be invited to participate a face-to-face semi-structured interview in order to explore their perceptions and opinions towards the strengths and limitations of the intervention(s) used, factors influencing the challenging behaviours of the disabled residents, and their suggested strategies in reducing their clients' challenging behaviours in their work setting.

ELIGIBILITY:
Inclusion Criteria:

* exhibiting at least one type of challenging behavior
* admitted at least 3 months for long-term care
* being dependent on nursing care and physical assistance in daily activities
* aged 18 to 64 years

Exclusion Criteria:

* seriously ill or completely bed-rest residents
* having infectious diseases
* frequently discharged to general hospital for acute care
* frequent home or day leave
* having pressure ulcer and/or severe contracture and deformity
* being restless and reluctant to stay in multisensory environment, or receive massage therapy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2013-04-15 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Behavior Problem Inventory (BPI-01): frequency and severity of challenging behaviours | Baseline (at recruitment)
  BPI-01 consists of 49 items with three subscales and has been widely employed in people with intellectual disability who are living in residential settings. This instrument is to evaluate the frequency and severity of challenging behaviours over the past two weeks of each assessment time points.
  Each item of the scale can be assessed on both frequency and severity of each kind of behaviour. The frequency scale is a 5-point rating scale: 0 - never, 1 - monthly, 2 - weekly, 3 - daily, and 4 - hourly. The severity scale is a 4-point Likert scale, denoted by: 0 - no problem, 1 - a slight problem, 2 - a moderate problem, and 3 - a severe problem. If a resident does not exhibit any behaviour listed in the item, "never" and "no problem" should be rated on that item.
Behavior Problem Inventory (BPI-01) | 5 weeks after intervention started (interim assessment)
  Behavior Problem Inventory (as described above) will be used to measure the frequency and severity of challenging behaviours by the end of week 5.
Behavior Problem Inventory (BPI-01) | 10 weeks after intervention started (Post-test 1)
  Behavior Problem Inventory (BPI-01) (as described above) will be used to measure the frequency and severity of challenging behaviours by the end of week 10.
Behavior Problem Inventory (BPI-01) | 12 weeks after intervention started (Post-test 2)
  Behavior Problem Inventory (as described above) will be used to measure the frequency and severity of challenging behaviours by the end of week 12.
Respiration and Pulse Rate | Baseline (at recruitment)
  Relaxation is a state of parasympathetic activation by vagal nerve, and suppressing the activity of sympathetic nervous system. If massage therapy and/or MSE indicate relaxation effect, the physiological parameters, i.e. pulse and respiration rates, are expected to drop to a lower level as compared with baseline readings after the interventions.
  Respiration rate and heart (pulse) rate will be measured 3 minutes just after the participants attended the intervention sessions. Their average values will be used for outcome analysis.
Respiration and Pulse Rate | 5 weeks after intervention started (interim assessment)
  Respiration rate and heart (pulse) rate will be measured 3 minutes just after the participants attended the intervention sessions by the end of week 5. Their average values will be used for outcome analysis.
Respiration and Pulse Rate | 10 weeks after intervention started (Post-test 1)
  Respiration rate and heart (pulse) rate will be measured 3 minutes just after the participants attended the intervention sessions by the end of week 10. Their average values will be used for outcome analysis.
Respiration and Pulse Rate | 12 weeks after intervention started (Post-test 2)
  Respiration rate and heart (pulse) rate will be measured 3 minutes by the end of week 12. Their average values will be used for outcome analysis.

SECONDARY OUTCOMES:
Alertness Observation Checklist (AOC) | Baseline (At recruitment)
  With the Alertness Observation Checklist (AOC), four levels of alertness of the participants can be distinguished: active, inactive and withdrawn, sleeping or drowsy, and agitated and discontented. Each level will be assigned with a color for presentation, including green for active level, orange for inactive and withdrawn state, red for sleepy or drowsy state, and blue for an agitated and discontented state. Frequency of alertness levels will be observed during the interventions. The averaged frequency is used for outcome analysis.
Alertness Observation Checklist (AOC) | 5 weeks after intervention started (interim assessment)
  Alertness Observation Checklist (AOC) will be used to measure the average amount of the four levels of alertness by the end of week 5.
Alertness Observation Checklist (AOC) | 10 weeks after intervention started (Post-test 1)
  Alertness Observation Checklist (AOC) will be used to measure the average amount of the four levels of alertness by the end of week 10.
Alertness Observation Checklist (AOC) | 12 weeks after intervention started (Post-test 2)
  Alertness Observation Checklist (AOC) will be used to measure the average amount of the four levels of alertness by the end of week 12.
Behaviour Checklist (BC) | Baseline (at recruitment)
  The Behaviour Checklist (BC) was developed by Shapiro et al. (1997) to assess the behavioral reactions toward multi-sensory environment and relevant psychological interventions. It consists of 22 items in which 16 items are for self-stimulating behaviours and 6 items for adaptive behaviours. Frequency of each of the listed behaviors in the checklist will be observed and counted at 1-minute intervals during the intervention sessions.
Behaviour Checklist (BC) | 5 weeks after intervention started (interim assessment)
  Behaviour Checklist (BC) will be used to measure the frequency of self-stimulating and adaptive behaviours by the end of week 5.
Behaviour Checklist (BC) | 10 weeks after intervention started (Post-test 1)
  Behaviour Checklist (BC) will be used to measure the frequency of self-stimulating and adaptive behaviours by the end of week 10.
Behaviour Checklist (BC) | 12 weeks after intervention started (Post-test 2)
  Behaviour Checklist (BC) will be used to measure the frequency of self-stimulating and adaptive behaviours by the end of week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Wai Tong CHIEN, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Siu Lam Hospital, Tuenmen, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chan JSL, Chien WT. A randomised controlled trial on evaluation of the clinical efficacy of massage therapy in a multisensory environment for residents with severe and profound intellectual disabilities: a pilot study. J Intellect Disabil Res. 2017 Jun;61(6):532-548. doi: 10.1111/jir.12377. Epub 2017 Apr 7. PMID 28387017